CLINICAL TRIAL: NCT04001738
Title: Evaluation of Direct Transfer to Angiography Suite vs. Computed Tomography Suite in Endovascular Treatment: Randomized Clinical Trial
Brief Title: Evaluation of Direct Transfer to Angiography Suite vs. Computed Tomography Suite in Endovascular Treatment: Randomized Clinical Trial (ANGIOCAT)
Acronym: ANGIOCAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Intermediate analysis
Sponsor: Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Manuel Requena Ruiz, Principal Investigator, Hospital Vall d'Hebron
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)156/2018
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Stroke, Acute
Keywords: Endovascular treatment; Large Vessel Occlusion
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct Transfer to Angio Suite (Active Comparator): After a fast neurological evaluation, patient will be direct transferred to angiography suite where endovascular treatment (EVT) team will be waiting for it. It will be done a cone beam-CT and if the image don't contraindicate endovascular treatment it will be performed and the large vessel occlusion will be confirmed by arteriography. If intravenous treatment have not been previously administered, it will be able to start in parallel.
  Interventions: Other: Direct Transfer to Angio Suite
- Direct Transfer to CT Scan (No Intervention): After a fast neurological evaluation, patient will be transferred to CT suite where usual image protocol will be performed (CT and CT-angio). Within 6 hours from onset CT perfusion could be required to take detections. Once interpreted image results, it will be decided intravenous and/or endovascular treatment.

INTERVENTIONS:
Other: Direct Transfer to Angio Suite — Patient will be direct transferred to angiography suite where EVT team will be waiting for it.
  Arms: Direct Transfer to Angio Suite

SUMMARY:
To evaluate the hypothesis that an ultra-fast triage with one-stop in angiography suite based on cone-beam CT compared to traditional protocol offers a better outcome in the distribution of the modified Rankin Scale scores at 90 days in acute ischemic stroke patients with suspected large vessel occlusion (LVO) within 6 hours from symptoms onset.

DETAILED DESCRIPTION:
Prospective, randomized, open, treatment-blinded trial of acute stroke patients with suspected large vessel occlusion within 6 hours from symptoms onset in which two strategies will be compared: Direct Transfer to Angiography Suite (DTAS) vs. Computed Tomography Suite (DTCT). The study will be unicentric however there is the possibility of incorporating new stroke centers with previous experience of at least 50 DTAS cases.

The RACE scale (Rapid Arterial oCclusion Evaluation) will be used as a prehospital screening tool to identify acute stroke patients with suspicion of LVO. Once prenotifying the imminent arrival and the verified inclusion and exclusion criteria by the Neurologist at arrival, the patient will be randomized by an app in one of both study protocols.

Subjects will be followed up to 90 days post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Large vessel occlusion suspected acute stroke codes (RACE>4) within 6 hours from stroke onset which are prenotified from emergency medical system.
* Confirmed NIHSS>10 at arrival.
* Good pre-stroke functional status (mRS≤2)
* Angiography suite available.
* Endovascular treatment team available (Neurologist, Interventionist, anesthesiologist, Nursery, Technicians…)

Exclusion Criteria:

* Hemodynamically unstable patients who requires of advanced vital support.
* Patients with an advanced disease that conditions a life expectancy lower than 6 months.
* Participation in other clinical trial with a drug or device which could influence in the outcome.
* Patients with neurological or psychiatric disease that could confound future evaluations.
* Lack of disponibility for 90 days tracing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-11-07 (Actual); Study Completion 2020-11-07 (Actual)

PRIMARY OUTCOMES:
Clinical outcome measurde by modified Rankin Scale score (shift analysis) | 90 days
  Modified Rankin Scale score in ischemic stroke patients with large vessel occlusion as evaluated through a structured telephone-based interview performed by a central assessor who is blinded to group assignment.
  Modified Rankin Scale measures functional status with a range from 0 (asymptomatic) to 6 (dead).
Rate of patients with treatment associated complications. | 72 hours
  Lack of treatment associated complications, mainly hemorrhagic transformation.

SECONDARY OUTCOMES:
Delay of inhospital times | 8 hours
  Time from door to groin puncture
Rate of dramatic improvement | 24 hours
  10 NIHSS points drop or NIHSS <2
Rate of good functional outcome | 90 days
  Modified Rankin Scale score ≤2
Rate of patients treated by endovascular treatment | 8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Vall d'Hebron University Hospital, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perez de la Ossa N, Carrera D, Gorchs M, Querol M, Millan M, Gomis M, Dorado L, Lopez-Cancio E, Hernandez-Perez M, Chicharro V, Escalada X, Jimenez X, Davalos A. Design and validation of a prehospital stroke scale to predict large arterial occlusion: the rapid arterial occlusion evaluation scale. Stroke. 2014 Jan;45(1):87-91. doi: 10.1161/STROKEAHA.113.003071. Epub 2013 Nov 26. PMID 24281224
- [Background] Ribo M, Boned S, Rubiera M, Tomasello A, Coscojuela P, Hernandez D, Pagola J, Juega J, Rodriguez N, Muchada M, Rodriguez-Luna D, Molina CA. Direct transfer to angiosuite to reduce door-to-puncture time in thrombectomy for acute stroke. J Neurointerv Surg. 2018 Mar;10(3):221-224. doi: 10.1136/neurintsurg-2017-013038. Epub 2017 Apr 26. PMID 28446535
- [Background] Jadhav AP, Kenmuir CL, Aghaebrahim A, Limaye K, Wechsler LR, Hammer MD, Starr MT, Molyneaux BJ, Rocha M, Guyette FX, Martin-Gill C, Ducruet AF, Gross BA, Jankowitz BT, Jovin TG. Interfacility Transfer Directly to the Neuroangiography Suite in Acute Ischemic Stroke Patients Undergoing Thrombectomy. Stroke. 2017 Jul;48(7):1884-1889. doi: 10.1161/STROKEAHA.117.016946. Epub 2017 May 23. PMID 28536177
- [Background] Psychogios MN, Behme D, Schregel K, Tsogkas I, Maier IL, Leyhe JR, Zapf A, Tran J, Bahr M, Liman J, Knauth M. One-Stop Management of Acute Stroke Patients: Minimizing Door-to-Reperfusion Times. Stroke. 2017 Nov;48(11):3152-3155. doi: 10.1161/STROKEAHA.117.018077. Epub 2017 Oct 10. PMID 29018132
- [Background] Mendez B, Requena M, Aires A, Martins N, Boned S, Rubiera M, Tomasello A, Coscojuela P, Muchada M, Rodriguez-Luna D, Rodriguez-Villatoro N, Juega J, Pagola J, Molina CA, Ribo M. Direct Transfer to Angio-Suite to Reduce Workflow Times and Increase Favorable Clinical Outcome. Stroke. 2018 Nov;49(11):2723-2727. doi: 10.1161/STROKEAHA.118.021989. PMID 30355182
- [Derived] Requena M, Olive-Gadea M, Muchada M, Hernandez D, Rubiera M, Boned S, Pinana C, Deck M, Garcia-Tornel A, Diaz-Silva H, Rodriguez-Villatoro N, Juega J, Rodriguez-Luna D, Pagola J, Molina C, Tomasello A, Ribo M. Direct to Angiography Suite Without Stopping for Computed Tomography Imaging for Patients With Acute Stroke: A Randomized Clinical Trial. JAMA Neurol. 2021 Sep 1;78(9):1099-1107. doi: 10.1001/jamaneurol.2021.2385. PMID 34338742